CLINICAL TRIAL: NCT06129448
Title: Evaluation of Tumor Necrosis Factor-alpha Levels and Cardiac Functions in Pediatric Patients Diagnosed With Type 1 Diabetes Mellitus
Brief Title: Tumor Necrosis Factor-alpha Levels and Cardiac Functions in Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Sirnak State Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Maze AYDEMIR, medical doctorat at pediatric cardiology unit, Sirnak State Hospital
Other Study IDs: Sirnakstatehospitalmaydemir001
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 1; Systolic Dysfunction; Diastolic Dysfunction
Keywords: systolic dysfunction; diastolic dysfunction; Diabetes mellitus type 1; pediatric; tissue doppler
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken for the analyses of TNF-a.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes Mellitus: We will include in this group patients with a diagnosis of T1DM, determined according to the World Health Organization criteria, who need insulin treatment and whose diabetes duration is more than 1 year. Patients will not have additional chronic diseases and will not have any other medical treatments other than insulin.
  Interventions: Diagnostic Test: transthoracic echocardiography
- Healthy Children: Patients will not have additional chronic diseases or other medical treatments. They will often be selected on a voluntary basis from patients who apply to pediatric cardiology with symptoms such as murmur or chest pain.
  Interventions: Diagnostic Test: transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: transthoracic echocardiography — All echocardiographic studies will be performed by one physician (Merve Maze AYDEMIR) using a commercially available echocardiographic system (P4-2 probe, DC-60, Mindray, Shenzhen, China) in the back-to-top or left lateral decubitus position. All images will be digitally stored from three cardiac cycles as standard apical four-chamber and parasternal short-axis views.

SUMMARY:
The goal of this clinical trial is to learn about the effect of type 1 diabetes mellitus on cardiac functions and evaluate the correlation of the dysfunction with the tumor necrosis factor-α (TNF-α) an inflammation-related factor. The study population will be the patients with the diagnosis of type 1 diabetes mellitus and the healthy children es the control group. The main question[s] it aims to answer are:

* Is diabetes affecting the systolic and diastolic cardiac functions
* Is diabetes affecting the left and the right ventricles equally?
* Does diabetes status, as assessed by HbA1c, have an impact on the occurrence of cardiac dysfunction?
* Is TNF-α can be a marker for early diagnosis of cardiac dysfunction? Diabetic patients will be examined by both a pediatric endocrinologist and a pediatric cardiologist. Transthoracic echocardiography will be performed and TNF-α will be evaluated for both the diabetic patients and the healthy children.

DETAILED DESCRIPTION:
Type 1 Diabetes Mellitus (T1DM) patients are at risk of developing cardiac dysfunction, a serious complication. Conventional echocardiography and tissue Doppler echocardiography are the most commonly used methods to evaluate cardiac functions. This study aims to prospectively assess the cardiac functions of pediatric patients diagnosed with T1DM. After routine pediatric endocrinology assessments, including anthropometric measurements, monitoring of blood glucose charts, and inquiring about complications related to diabetes, patients will be referred for pediatric cardiology evaluation. Standard pediatric cardiac examination, electrocardiographic evaluation, and echocardiography, including conventional transthoracic echocardiography and tissue Doppler echocardiography, will be performed.

Patients with a T1DM diagnosis typically provide blood samples for standard tests (HgA1c, blood glucose, routine biochemistry, etc.) following each pediatric endocrinology visit. In this study, an additional blood sample will be taken during blood collection to measure tumor necrosis factor-alpha (TNF-α) levels. Previous studies have shown elevated TNF-α levels in T1DM patients. This study aims to investigate its potential impact on cardiac function. Similarly, an age- and gender-matched control group of healthy children without T1DM will be established. This control group will also undergo echocardiographic evaluation, and TNF-α levels in their blood will be measured. Subsequently, statistical analysis will be conducted.

Through these assessments, this study aims to determine whether there is a deterioration in systolic and diastolic heart functions in the pediatric T1DM patient group compared to the control group and to evaluate the effect of TNF-α levels on these results.

ELIGIBILITY:
Inclusion Criteria:

-Patients with a diagnosis of Type 1 Diabetes Mellitus (T1DM) who have been under follow-up for at least 1 year (for the patient group)

Exclusion Criteria:

* Having an additional cardiac anomaly
* Having an additional chronic medical condition

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with a diagnosis of Type 1 Diabetes Mellitus (T1DM) for more than 1 year will be the first group.
  The second group will consist of healthy children without any additional medical conditions, who are similar in terms of age and gender to the children in the first group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
The percentage of T1DM patients who had decreased systolic left ventricle functions. | 1 month
  We will include Type 1 DM patients diagnosed for over a year. After routine pediatric endocrinology assessments, they'll visit the pediatric cardiology clinic. By echocardiography, ejection fraction (EF) and fractional shortening (FS) will be measured in percentages. For these calculations, Left ventricular end-diastolic dimension, Interventricular septum, and LV posterior wall thickness in systole and diastole will be measured in mm. The expected normal value for EF is >%55 and FS > %30.
The percentage of T1DM patients who had decreased diastolic left ventricle functions. | 1 month
  To assess diastolic dysfunction by echocardiography, the mitral diastolic flow tracings will be imaged in pulsed Doppler with sample volume sited at the tips of the mitral leaflets. Peak velocities of early (E) and late (A) filling (m/s) will be derived from atrioventricular valve inflow velocity profiles. The early to late peak velocities (E/A) ratio will be calculated. In addition, by tissue Doppler imaging echocardiography, myocardial wall motion velocity will be recorded by activating the pulsed-wave (PW) tissue Doppler function on the same machine. LV septal and lateral mitral annulus measures: early (Em) and late (Am) (m/s) diastolic myocardial velocities, isovolumic contraction time , isovolumic relaxation time and ejection time (ms) will be measured. The myocardial performance index will be calculated as (IVCT + IVRT)/ET.
The percentage of T1DM patients who had decreased right ventricle functions. | 1 month
  The tricuspid diastolic flow tracings will be imaged in pulsed Doppler to assess diastolic dysfunction by echocardiography. Peak velocities of early (E) and late (A) filling (m/s) will be derived from atrioventricular valve inflow velocity profiles. The early to late peak velocities (E/A) ratio will be calculated. In addition, by tissue. For lateral tricuspid annulus, early (Em) and late (Am) (m/s) diastolic myocardial velocities, isovolumic contraction time, isovolumic relaxation time, and ejection time (ms) will be measured by Doppler imaging echocardiography. The myocardial performance index will be calculated as (IVCT + IVRT)/ET. Tricuspid annular plane systolic excursion (TAPSE) (mm) will be assessed for systolic function.
Effect of Tumor necrosis factor- α (TNF-α) on cardiac functions | 1 month
  This study will include T1DM patients diagnosed for over a year who have undergone routine pediatric endocrinology evaluations. We'll collect extra blood samples to measure TNF-α levels (pg/mL). We will evaluate whether blood TNF-α levels are higher in patients who develop systolic and/or diastolic dysfunction compared to patients who do not develop dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE MA AYDEMİR, Study Director — Sirnak State Hospital; Tahir Çağdaş, Principal Investigator — Sirnak State Hospital; Özge Doğan, Principal Investigator — Sirnak State Hospital; Veysel Tahiroğlu, Principal Investigator — Şırnak Üniversitesi; Cem Mete, Principal Investigator — Sirnak State Hospital; Hasan Karageçili, Principal Investigator — Siirt University
Locations (1):
- Sirnak State Hospital, Şırnak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoldas T, Orun UA, Sagsak E, Aycan Z, Kaya O, Ozgur S, Karademir S. Subclinical left ventricular systolic and diastolic dysfunction in type 1 diabetic children and adolescents with good metabolic control. Echocardiography. 2018 Feb;35(2):227-233. doi: 10.1111/echo.13764. Epub 2017 Dec 3. PMID 29205484
- [Background] M Abd-El Aziz F, Abdelghaffar S, M Hussien E, M Fattouh A. Evaluation of Cardiac Functions in Children and Adolescents with Type 1 Diabetes. J Cardiovasc Ultrasound. 2017 Mar;25(1):12-19. doi: 10.4250/jcu.2017.25.1.12. Epub 2017 Mar 27. PMID 28400931
- [Background] Dos Santos Haber JF, Barbalho SM, Sgarbi JA, de Argollo Haber RS, de Labio RW, Laurindo LF, Chagas EFB, Payao SLM. The Relationship between Type 1 Diabetes Mellitus, TNF-alpha, and IL-10 Gene Expression. Biomedicines. 2023 Apr 7;11(4):1120. doi: 10.3390/biomedicines11041120. PMID 37189738